CLINICAL TRIAL: NCT04799132
Title: Association Between Body Mass Index and High-flow Cannula Therapy Success in Patients With Severe Covid 19 Related Pneumonia. Retrospective Study.
Brief Title: Association Between Body Mass Index and HFNC Therapy Success
Status: Completed | Type: Observational
Sponsor: Clínica del country (Other)
Responsible Party: Principal Investigator, Carlos Augusto Celemín Florez, MD., Principal Investigator., Clínica del country
Other Study IDs: BMI AND HFNC
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Obesity; Overweight; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Obesity; Overweight; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients over 18 years of age who are admitted to the Intermediate Care Unit of the Clinica del Country and the Clinica la Colina, with symptoms suggestive of severe pneumonia secondary to COVID-19 infection and acute hypoxemic respiratory failure. The primary outcome will be to determine the relationship between body mass index and high-flow cannula therapy success defined as: No need for mechanical ventilation.

DETAILED DESCRIPTION:
All adult patients over 18 years of age admitted to the intermediate care service of the participating center with suspected SARS-CoV-2 pneumonia will be considered as potential candidates for the study.

The medical records of patients in our cohort who require high-flow cannula therapy and who met all the inclusion criteria and none of the exclusion criteria will be reviewed.All data will be processed and analyzed using the SPSS 26 software once the study is completed. study sample

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age.
2. Diagnosis of severe pneumonia secondary to COVID-19 infection and acute respiratory distress syndrome, defined by upper and lower respiratory symptoms plus positive C-reactive protein test for COVID-19.
3. Patient admission to the Clinical del Country and Clinica de la Colina intermediate care units.
4. Oxygen therapy by high-flow system (high-flow cannula) requirement.
5. Anthropometric data availability upon admission to our facilities.

Exclusion Criteria:

1. Patients with a survival expectancy of less than 12 months according to the Charlson scale categorization or patients with oncological pathology.
2. Patients under 18 years of age.
3. Pregnant women.
4. Patients with cardiogenic pulmonary edema.
5. History of chronic liver disease or cirrhosis Child - Pugh C.
6. Patients with contraindications to high-flow cannula therapy initiation.
7. Patients with respiratory, hemodynamic and neurological indications that contraindicate HFNC initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who are admitted to the Intermediate Care Unit of the Clinica del Country and the Clinica la Colina, with symptoms suggestive of severe pneumonia secondary to COVID-19 infection and acute hypoxemic respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 1 year.
  To determine the relationship between body mass index "BMI" calculated by kg / m2 (BMI was classified in the following categories: normal weight: 18.5-24.9 kg / m2, overweight: 25-29.9 kg / m2, and obesity: ≥ 30 kg / m2) and high-flow cannula therapy success defined as: No need for mechanical ventilation.

SECONDARY OUTCOMES:
Demographic and laboratory characteristics | 1 year
  Describe the clinical, demographic and laboratory characteristics in a population of 303 patients in Bogotá, Colombia with severe pneumonia defined by ATS criteria (confusion, urea >7 mmol/L, respiratory rate ≥30 min-1, low blood pressure, and age ≥65 years) score except age, arterial oxygen pressure/fraction inspired oxygen (PaO2/FiO2) ≤250 mmHg, multilobar infiltrates, leucopenia, thrombocytopenia, and hypothermia.) secondary to COVID 19 infection (positive C-Reactive protein) and acute hypoxemic respiratory failure defined by a PaFio2 < 300, in the intermediate care service of the Clínica del Country and Clínica La Colina, between March 2020 and March 2021.
Body mass index as a predictor | 1 year
  Evaluate the body mass index as a predictor of success in high-flow cannula therapy.
Body mass index and HFNC success | 1 year
  Evaluate the relationship between body mass index and high-flow nasal cannula therapy success.
Mortality | 1 year
  Describe the mortality of patients with high-flow cannula therapy in our medical facilities.
Hospital stay. | 1 year
  The relationship between hospital stay (days) and body mass index in our patients' cohort will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica del Country., Bogotá, Colombia

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] de Frel DL, Atsma DE, Pijl H, Seidell JC, Leenen PJM, Dik WA, van Rossum EFC. The Impact of Obesity and Lifestyle on the Immune System and Susceptibility to Infections Such as COVID-19. Front Nutr. 2020 Nov 19;7:597600. doi: 10.3389/fnut.2020.597600. eCollection 2020. PMID 33330597
- [Background] Rochwerg B, Einav S, Chaudhuri D, Mancebo J, Mauri T, Helviz Y, Goligher EC, Jaber S, Ricard JD, Rittayamai N, Roca O, Antonelli M, Maggiore SM, Demoule A, Hodgson CL, Mercat A, Wilcox ME, Granton D, Wang D, Azoulay E, Ouanes-Besbes L, Cinnella G, Rauseo M, Carvalho C, Dessap-Mekontso A, Fraser J, Frat JP, Gomersall C, Grasselli G, Hernandez G, Jog S, Pesenti A, Riviello ED, Slutsky AS, Stapleton RD, Talmor D, Thille AW, Brochard L, Burns KEA. The role for high flow nasal cannula as a respiratory support strategy in adults: a clinical practice guideline. Intensive Care Med. 2020 Dec;46(12):2226-2237. doi: 10.1007/s00134-020-06312-y. Epub 2020 Nov 17. PMID 33201321
- [Background] Smati S, Tramunt B, Wargny M, Caussy C, Gaborit B, Vatier C, Verges B, Ancelle D, Amadou C, Bachir LA, Bourron O, Coffin-Boutreux C, Barraud S, Dorange A, Fremy B, Gautier JF, Germain N, Larger E, Laugier-Robiolle S, Meyer L, Monier A, Moura I, Potier L, Sabbah N, Seret-Begue D, Winiszewski P, Pichelin M, Saulnier PJ, Hadjadj S, Cariou B, Gourdy P; CORONADO investigators. Relationship between obesity and severe COVID-19 outcomes in patients with type 2 diabetes: Results from the CORONADO study. Diabetes Obes Metab. 2021 Feb;23(2):391-403. doi: 10.1111/dom.14228. Epub 2020 Nov 6. PMID 33051976
- [Background] Magdy Beshbishy A, Hetta HF, Hussein DE, Saati AA, C Uba C, Rivero-Perez N, Zaragoza-Bastida A, Shah MA, Behl T, Batiha GE. Factors Associated with Increased Morbidity and Mortality of Obese and Overweight COVID-19 Patients. Biology (Basel). 2020 Sep 9;9(9):280. doi: 10.3390/biology9090280. PMID 32916925
- [Background] Xia J, Zhang Y, Ni L, Chen L, Zhou C, Gao C, Wu X, Duan J, Xie J, Guo Q, Zhao J, Hu Y, Cheng Z, Zhan Q. High-Flow Nasal Oxygen in Coronavirus Disease 2019 Patients With Acute Hypoxemic Respiratory Failure: A Multicenter, Retrospective Cohort Study. Crit Care Med. 2020 Nov;48(11):e1079-e1086. doi: 10.1097/CCM.0000000000004558. PMID 32826432
- [Background] Petrakis D, Margina D, Tsarouhas K, Tekos F, Stan M, Nikitovic D, Kouretas D, Spandidos DA, Tsatsakis A. Obesity - a risk factor for increased COVID-19 prevalence, severity and lethality (Review). Mol Med Rep. 2020 Jul;22(1):9-19. doi: 10.3892/mmr.2020.11127. Epub 2020 May 5. PMID 32377709
- [Background] Popkin BM, Du S, Green WD, Beck MA, Algaith T, Herbst CH, Alsukait RF, Alluhidan M, Alazemi N, Shekar M. Individuals with obesity and COVID-19: A global perspective on the epidemiology and biological relationships. Obes Rev. 2020 Nov;21(11):e13128. doi: 10.1111/obr.13128. Epub 2020 Aug 26. PMID 32845580
- [Background] Sales-Peres SHC, de Azevedo-Silva LJ, Bonato RCS, Sales-Peres MC, Pinto ACDS, Santiago Junior JF. Coronavirus (SARS-CoV-2) and the risk of obesity for critically illness and ICU admitted: Meta-analysis of the epidemiological evidence. Obes Res Clin Pract. 2020 Sep-Oct;14(5):389-397. doi: 10.1016/j.orcp.2020.07.007. Epub 2020 Aug 3. PMID 32773297
- [Background] Cummings MJ, Baldwin MR, Abrams D, Jacobson SD, Meyer BJ, Balough EM, Aaron JG, Claassen J, Rabbani LE, Hastie J, Hochman BR, Salazar-Schicchi J, Yip NH, Brodie D, O'Donnell MR. Epidemiology, clinical course, and outcomes of critically ill adults with COVID-19 in New York City: a prospective cohort study. Lancet. 2020 Jun 6;395(10239):1763-1770. doi: 10.1016/S0140-6736(20)31189-2. Epub 2020 May 19. PMID 32442528
- [Background] Nogueira-de-Almeida CA, Del Ciampo LA, Ferraz IS, Del Ciampo IRL, Contini AA, Ued FDV. COVID-19 and obesity in childhood and adolescence: a clinical review. J Pediatr (Rio J). 2020 Sep-Oct;96(5):546-558. doi: 10.1016/j.jped.2020.07.001. Epub 2020 Aug 4. PMID 32768388
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Contou D, Cally R, Sarfati F, Desaint P, Fraisse M, Plantefeve G. Causes and timing of death in critically ill COVID-19 patients. Crit Care. 2021 Feb 23;25(1):79. doi: 10.1186/s13054-021-03492-x. No abstract available. PMID 33622349
- [Background] Dale CR, Starcher RW, Chang SC, Robicsek A, Parsons G, Goldman JD, Vovan A, Hotchkin D, Gluckman TJ. Surge effects and survival to hospital discharge in critical care patients with COVID-19 during the early pandemic: a cohort study. Crit Care. 2021 Feb 17;25(1):70. doi: 10.1186/s13054-021-03504-w. PMID 33596975
- [Background] Williamson EJ, Walker AJ, Bhaskaran K, Bacon S, Bates C, Morton CE, Curtis HJ, Mehrkar A, Evans D, Inglesby P, Cockburn J, McDonald HI, MacKenna B, Tomlinson L, Douglas IJ, Rentsch CT, Mathur R, Wong AYS, Grieve R, Harrison D, Forbes H, Schultze A, Croker R, Parry J, Hester F, Harper S, Perera R, Evans SJW, Smeeth L, Goldacre B. Factors associated with COVID-19-related death using OpenSAFELY. Nature. 2020 Aug;584(7821):430-436. doi: 10.1038/s41586-020-2521-4. Epub 2020 Jul 8. PMID 32640463
- [Background] Kompaniyets L, Goodman AB, Belay B, Freedman DS, Sucosky MS, Lange SJ, Gundlapalli AV, Boehmer TK, Blanck HM. Body Mass Index and Risk for COVID-19-Related Hospitalization, Intensive Care Unit Admission, Invasive Mechanical Ventilation, and Death - United States, March-December 2020. MMWR Morb Mortal Wkly Rep. 2021 Mar 12;70(10):355-361. doi: 10.15585/mmwr.mm7010e4. PMID 33705371